CLINICAL TRIAL: NCT04933942
Title: Romiplostim for Thrombocytopenia Induced by Lomustine at First Progression of MGMT Promoter-methylated Glioblastoma: a Randomized Phase II Open Label Multicenter Study
Brief Title: Phase II Trial of Romiplostim for Thrombocytopenia Induced by Lomustine at First Progression of MGMT Promoter-meth Glioblastoma
Acronym: RIGOLETTO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Amgen withdrew interest in providing further financial support
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1926-BTG
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: First Progression of MGMT Promoter-methylated Glioblastoma
Keywords: First progression; MGMT promoter-methylated glioblastoma; Phase II; Romiplostim; Lomustine
MeSH Terms: interventions — Lomustine; romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Lomustine alone
  Interventions: Drug: Lomustine
- Experimental group (Experimental): Lomustine plus Romiplostim
  Interventions: Drug: Lomustine; Drug: Romiplostim

INTERVENTIONS:
Drug: Lomustine — Oral administration of Lomustine
Drug: Romiplostim — Subcutaneous administration of Romiplostim
  Arms: Experimental group

SUMMARY:
Romiplostim for low platelets caused by lomustine chemotherapy in patients with first recurrence (growing back) of a brain tumor, glioblastoma that is MGMT methylated.

Lomustine is an anticancer drug often used to treat glioblastoma that grows back after initial treatment. This anticancer drug can cause side effects. The most frequent and potentially serious side effect of all is lowering of the blood platelets. Low platelets can cause bleedings in the the stomach and intestines, the skin, the brain and other systems and tissues.

Low platelets are also the main cause of delaying or prematurely (ending treatment before the planned end) stopping chemotherapy. There is no treatment for low platelets except platelet transfusions. Romiplostim is a drug that stimulates the production of platelets in the bone marrow. It is an approved drug in USA, Europe, Australia and Switzerland for a special type of blood disease in which the body breaks down its own blood platelets.

The purpose of the study is to start the treatment with romiplostim once low platelets are diagnosed in order to restore the platelet count and to prevent the platelet count from dropping again during the lomustine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more on day of signing informed consent
* Karnofsky Performance Score (KPS) of 60-100
* Life expectancy > 8 weeks
* Stable or decreasing dose of steroids for at least 1 week prior to enrolment
* Glioblastoma isocitrate dehydrogenase (IDH1) R132H wild-type, per cIMPACT NOW recommendations (Brat et al., 2018; Brat et al., 2020)
* MGMT promoter methylation determined by methylation-specific PCR or pyrosequencing or methylation profiling per local assessment.
* Treatment with lomustine alone for first progression after any treatment comprising intent to treat with standard TMZ /RT →TMZ for newly diagnosed glioblastoma, with at least one dose of maintenance TMZ received. Hypofractionated regimens of RT are allowed. Patients should have received at least 75% of the RT dose. Patients enrolled in a clinical study for newly diagnosed glioblastoma and treated with standard of care and an experimental agent can participate. Patients who had RT alone or TMZ alone for newly diagnosed glioblastoma are not eligible. Patients must have received at least one dose of lomustine
* Clinically relevant thrombocytopenia defined as thrombocytopenia requiring dose delay of lomustine for at least one week (more than 7 days) (for any grade of toxicity) or requiring a dose reduction of lomustine because of grade 3 or 4 thrombocytopenia
* Diagnosis of first progression according to RANO criteria (Wen et al., 2010) more than 3 months after the end of radiotherapy for first-line treatment
* Patients may have been operated for recurrence. If operated, patients should have fully recovered from surgery as assessed by the investigator. Criteria for full recovery include absence of post-operative infection, recovery from medical complications (CTCAE grade 0 and 1 acceptable). Residual and measurable disease after surgery is not required, but surgery must have confirmed the recurrence. The post-surgery MRI (performed within 72 h) can be used for enrolment if dated within 6 weeks of enrolment.
* For non-operated patients: recurrent disease must correspond to at least one bi-dimensionally measurable contrast-enhancing lesion with clearly defined margins by MRI scan, with minimal diameters of 10 mm (10x10 mm), visible on 2 or more axial slices 5 mm apart (measurable disease according to RANO criteria). The MRI can be used for enrolment if dated within 6 weeks prior to enrolment.
* In case of clinical deterioration or increase of steroids since the last MRI, a new MRI should be done prior to enrolment and should be dated within 6 weeks prior to enrolment.
* Patients diagnosed with a venous thromboembolism or thrombotic events within the last 3 months can be enrolled if they have been on a stable regimen of anticoagulants for at least 14 days.
* Capacity for adequate fluid and oral intake
* Adequate bone marrow (except for platelet count, which can be <100 x 109/L at enrolment), renal and hepatic function within 7 days before enrolment
* Hemoglobin ≥ 8 g/dl
* Leukocytes count NOT requiring CGSF per local Standard of Care
* Total bilirubin ≤ 1.5 ULN
* Alanine transaminase (ALT), Aspartate Transaminase (AST), alkaline phosphatase (ALP) ≤ 2.5 × ULN
* Serum creatinine < 1.5 x ULN or creatinine clearance (CrCl) > 30 mL/min (using the Cockcroft-Gault formula)
* Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test within 7 days prior to enrolment.
* Patients of childbearing / reproductive potential must agree to use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 6 months after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly (see Appendix G)
* Patients must also agree not to donate sperm during the study and for 6 months after receiving the last dose of study treatment
* Women who are breast feeding must agree to discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment
* Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments
* Before patient enrolment, written informed consent must be given according to ICH/GCP, and national/local regulations

Exclusion Criteria:

* Radiotherapy or stereotactic radiosurgery for the treatment of first progression prior to enrolment in this study
* Known further progression after initiation of lomustine at the time of enrolment. Any suspicion of progression should be explored by a new MRI prior to enrolment
* Prior exposure to romiplostim or other thrombopoietin (TPO) mimetics
* Other hematological toxicity (anemia, neutropenia) requiring erythropoietin or GCSF
* Contraindications for MRI, including intolerance of gadolinium as a contrast agent
* Known coagulation disease or known hematological disease even if resolved.
* Known hypercoagulative state (e.g., factor V Leiden, ATIII deficiency, protein C deficiency, protein S deficiency, antiphospholipid antibody syndrome)
* Clinically significant cardiac comorbidities, including: history of arterial thrombotic events (e.g., myocardial ischemia, transient ischemic attack, or stroke) within 6 months prior to screening, any history of active congestive heart failure (NYHA class II to IV), symptomatic ischaemia, including myocardial infarction, uncontrolled cardiac arrythmias, clinically significant ECG abnormalities, including screening ECG with QTc interval > 470 msec in women, > 450 msec in men, known pericardial disorder.
* History or present acute lymphoblastic leukaemia, acute myeloid leukaemia, any myeloid malignancy, myelodysplastic syndrome, myeloproliferative disease, multiple myeloma
* Evidence of active infection within 2 weeks prior to enrolment
* Known hypersensitivity to any E-coli derived product
* Known hypersensitivity to the active substances or to any of the excipients of the study drugs
* Any live attenuated vaccines, such as yellow fever vaccine, within the last 3 months before lomustine initiation.
* Known coeliac disease or wheat allergy
* Concurrent severe or uncontrolled medical disease (e.g., active systemic infection, diabetes, hypertension, coronary artery disease) that, in the opinion of the Investigator, would compromise the safety of the patient or compromise the ability of the patient to complete the study
* Known human immunodeficiency virus infection or acquired immune deficiency syndrome
* Known chronic active HBV or HCV within 4 months prior to enrolment
* Previous other malignancies, except for any previous malignancy which was treated with curative intent more than 2 years prior to enrolment, and except for adequately controlled limited basal cell carcinoma of the skin, adequately treated and without evidence of disease non-melanoma of the skin, squamous carcinoma of the skin and carcinoma in situ of the cervix, adequately treated breast ductal carcinoma in situ without evidence of disease, prostatic intraepithelial neoplasia without evidence of prostate cancer. Low risk prostate cancer (cT1-2a N0 and Gleason score ≤ 6 and PSA < 10 ng/mL), either totally resected or irradiated with curative intent (with PSA of less than or equal to 0.1 ng/mL) or under active surveillance as per ESMO guidelines
* Pregnant women
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 5 months after the last patient in

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 months after the last patient in
the Health-related Quality of Life (HRQoL) | 5 months after the last patient in
  HRQoL will be assessed with the EORTC Quality of Life Questionnaire (QLQ-C30) version 3.
Frequency of worst Adverse Events (AEs) | 5 months after the last patient in
  This study will use the International Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, for adverse event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Le Rhun, Principal Investigator — EORTC Study Coordinator
Locations (5):
- Spain (3):
  - Hospital Clinic Universitari de Barcelona, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
- Switzerland (2):
  - Oncology Institute of Southern Switzerland, Bellinzona
  - UniversitaetsSpital, Zurich